CLINICAL TRIAL: NCT02578355
Title: National Plaque Registry and Database
Acronym: OPeRA
Status: Not yet recruiting | Type: Observational
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: Hungarian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Pál Maurovich-Horvat, Assistant Professor, Semmelweis University Heart and Vascular Center
Other Study IDs: The OPeRA study
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Atherosclerosis; Coronary Artery Disease; Cardiovascular Disease
Keywords: Atherosclerosis; Coronary Artery Disease; Cardiovascular Disease; Coronary Computed Tomographic Angiography; CCTA; Myocardial Infarction; MI; OPeRA
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Cardiovascular Diseases; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coronary CT Angiography (CCTA): Patients included in the OPeRA Registry are those that have previously undergone clinically-indicated CCTA as part of their standard of care.

SUMMARY:
The ultimate goal of this project is to develop a risk score to identify patients with vulnerable coronary atherosclerotic plaques, who are prone to suffer acute coronary syndrome. Early identification of vulnerable plaques may have an enormous impact on public health through primary and secondary prevention of acute myocardial infarction.

Investigators hypothesize that a risk score that incorporates non-invasive coronary CT imaging (calcium score and/or coronary CTA) in combination with clinical characteristics (classical risk prediction models) will improve the identification of patients who are at highest risk to suffer myocardial infarction or sudden cardiac death.

The overall goal of the OPeRA project is to develop, implement and validate a novel risk assessment tool based on image markers and clinical characteristics to identify patients who are at increased risk to suffer myocardial infarction or sudden cardiac death.

DETAILED DESCRIPTION:
The primary goals of OPeRA consortium:

To develop a national coronary CTA registry with the collaboration of all major cardiac CT centers of Hungary (Országos Plaque Regiszter és Adatbázis - NatiOnal Plaque Registry and DAtabase, OPeRA).

1. To develop a novel risk assessment tool (OPeRA score) based on image markers and clinical characteristics.
2. To identify and validate novel vulnerable coronary plaque image markers and assess their prognostic value.

Secondary goals:

1. To develop a standardized and structured, national coronary CTA reporting system.
2. To establish a national quality control system that monitors the quantity of iodinated contrast agent and the patients' radiation dose.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Subject providing written informed consent
* Scheduled to undergo a clinically indicated coronary CTA

Exclusion Criteria:

* Age <18 years
* Suspicion of acute coronary syndrome (acute myocardial infarction and unstable angina)
* Recent prior myocardial infarction within 30 days prior to coronary CTA or between coronary CTA and ICA
* Pregnancy or unknown pregnancy status in subject of childbearing potential
* Subject requires an emergent procedure
* Evidence of ongoing or active clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure with systolic blood pressure <90 mmHg, and severe congestive heart failure (NYHA III or IV) or acute pulmonary edema
* Inability to comply with study procedures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent clinically indicated coronary CTA are involved in the sudy.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2016-09; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
All cause death | 10 years

SECONDARY OUTCOMES:
Myocardial infarction | 10 years
Unstable angina | 10 years
Target vessel revascularization | 10 years
CAD-related hospitalization | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Pál Maurovich-Horvat, MD, PhD, MPH, Principal Investigator — Heart and Vascular Center, Smellweis University
Locations (11):
- Hungary (11):
  - University of Pécs, Pécs, Baranya
  - Pándy Kálmán County Hospital, Gyula, Bekes County
  - Borsod-Abaúj-Zemplén County Hospital and Teaching Hospital, Miskolc, Borsod-Abaúj-Zenpén
  - University of Szeged, Szeged, Csongrád megye
  - Petz Aladár County Teaching Hospital, Győr, Győr-Moson-Sopron
  - University of Debrecen, Debrecen, Hajdú-Bihar
  - Markhot Ferenc Teaching Hospital and Clinic, Eger, Heves County
  - Homeland Defence Hospital, Budapest, Pest County
  - Health Centrum, Kaposvár University, Kaposvár, Somogy County
  - Markusovszky Teaching Hospital, Szombathely, Vas County
  - Pozitron Diagnostic Center, Budapest

REFERENCES:
- [Background] Nichols M, Townsend N, Scarborough P, Rayner M. Cardiovascular disease in Europe: epidemiological update. Eur Heart J. 2013 Oct;34(39):3028-34. doi: 10.1093/eurheartj/eht356. Epub 2013 Sep 7. PMID 24014390
- [Background] Narula J, Strauss HW. The popcorn plaques. Nat Med. 2007 May;13(5):532-4. doi: 10.1038/nm0507-532. No abstract available. PMID 17479093
- [Background] Braunwald E. Epilogue: what do clinicians expect from imagers? J Am Coll Cardiol. 2006 Apr 18;47(8 Suppl):C101-3. doi: 10.1016/j.jacc.2005.10.072. No abstract available. PMID 16631504
- [Background] Goff DC Jr, Lloyd-Jones DM, Bennett G, Coady S, D'Agostino RB, Gibbons R, Greenland P, Lackland DT, Levy D, O'Donnell CJ, Robinson JG, Schwartz JS, Shero ST, Smith SC Jr, Sorlie P, Stone NJ, Wilson PW, Jordan HS, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the assessment of cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S49-73. doi: 10.1161/01.cir.0000437741.48606.98. Epub 2013 Nov 12. No abstract available. PMID 24222018
- [Background] Genders TS, Steyerberg EW, Hunink MG, Nieman K, Galema TW, Mollet NR, de Feyter PJ, Krestin GP, Alkadhi H, Leschka S, Desbiolles L, Meijs MF, Cramer MJ, Knuuti J, Kajander S, Bogaert J, Goetschalckx K, Cademartiri F, Maffei E, Martini C, Seitun S, Aldrovandi A, Wildermuth S, Stinn B, Fornaro J, Feuchtner G, De Zordo T, Auer T, Plank F, Friedrich G, Pugliese F, Petersen SE, Davies LC, Schoepf UJ, Rowe GW, van Mieghem CA, van Driessche L, Sinitsyn V, Gopalan D, Nikolaou K, Bamberg F, Cury RC, Battle J, Maurovich-Horvat P, Bartykowszki A, Merkely B, Becker D, Hadamitzky M, Hausleiter J, Dewey M, Zimmermann E, Laule M. Prediction model to estimate presence of coronary artery disease: retrospective pooled analysis of existing cohorts. BMJ. 2012 Jun 12;344:e3485. doi: 10.1136/bmj.e3485. PMID 22692650
- [Background] Libby P. Mechanisms of acute coronary syndromes and their implications for therapy. N Engl J Med. 2013 May 23;368(21):2004-13. doi: 10.1056/NEJMra1216063. No abstract available. PMID 23697515
- [Background] Virmani R, Kolodgie FD, Burke AP, Farb A, Schwartz SM. Lessons from sudden coronary death: a comprehensive morphological classification scheme for atherosclerotic lesions. Arterioscler Thromb Vasc Biol. 2000 May;20(5):1262-75. doi: 10.1161/01.atv.20.5.1262. No abstract available. PMID 10807742
- [Background] Narula J, Garg P, Achenbach S, Motoyama S, Virmani R, Strauss HW. Arithmetic of vulnerable plaques for noninvasive imaging. Nat Clin Pract Cardiovasc Med. 2008 Aug;5 Suppl 2:S2-10. doi: 10.1038/ncpcardio1247. PMID 18641603
- [Background] Maurovich-Horvat P, Ferencik M, Voros S, Merkely B, Hoffmann U. Comprehensive plaque assessment by coronary CT angiography. Nat Rev Cardiol. 2014 Jul;11(7):390-402. doi: 10.1038/nrcardio.2014.60. Epub 2014 Apr 22. PMID 24755916
- [Background] Falk E, Nakano M, Bentzon JF, Finn AV, Virmani R. Update on acute coronary syndromes: the pathologists' view. Eur Heart J. 2013 Mar;34(10):719-28. doi: 10.1093/eurheartj/ehs411. Epub 2012 Dec 13. PMID 23242196
- [Background] Maurovich-Horvat P, Ferencik M, Bamberg F, Hoffmann U. Methods of plaque quantification and characterization by cardiac computed tomography. J Cardiovasc Comput Tomogr. 2009 Nov-Dec;3 Suppl 2:S91-8. doi: 10.1016/j.jcct.2009.10.012. Epub 2009 Oct 31. PMID 20129522
- [Background] Leipsic J, Abbara S, Achenbach S, Cury R, Earls JP, Mancini GJ, Nieman K, Pontone G, Raff GL. SCCT guidelines for the interpretation and reporting of coronary CT angiography: a report of the Society of Cardiovascular Computed Tomography Guidelines Committee. J Cardiovasc Comput Tomogr. 2014 Sep-Oct;8(5):342-58. doi: 10.1016/j.jcct.2014.07.003. Epub 2014 Jul 24. No abstract available. PMID 25301040
- [Background] Maurovich-Horvat P, Hoffmann U, Vorpahl M, Nakano M, Virmani R, Alkadhi H. The napkin-ring sign: CT signature of high-risk coronary plaques? JACC Cardiovasc Imaging. 2010 Apr;3(4):440-4. doi: 10.1016/j.jcmg.2010.02.003. No abstract available. PMID 20394906
- [Background] Engel LC, Lee AM, Seifarth H, Sidhu MS, Brady TJ, Hoffmann U, Ghoshhajra BB. Weekly dose reports: the effects of a continuous quality improvement initiative on coronary computed tomography angiography radiation doses at a tertiary medical center. Acad Radiol. 2013 Aug;20(8):1015-23. doi: 10.1016/j.acra.2013.04.012. PMID 23830607